CLINICAL TRIAL: NCT02177422
Title: Open-Label Follow-up Trial on Efficacy and Safety of Chronic Administration of Telmisartan 80 mg (Micardis®) Tablets as Monotherapy or in Combination With Hydrochlorothiazide or Other Antihypertensive Medications in Patients With Mild to Moderate Hypertension
Brief Title: Efficacy and Safety of Chronic Administration of Telmisartan as Monotherapy or in Combination With Hydrochlorothiazide or Other Antihypertensive Medications in Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.260
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

ARMS (1):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan — telmisartan 80 mg once daily
Drug: Hydrochlorothiazide — 12.5 mg or 25 mg Hydrochlorothiazide in addition to telmisartan in case that the goal response (mean sitting diastolic blood pressure < 90 mmHg) is not met after at least 4 weeks of treatment with telmisartan

SUMMARY:
The primary objective of this trial was to assess the efficacy and safety of telmisartan 80 mg during open-label, long-term treatment. An additional objective was to assess the efficacy and safety of concomitant administration of telmisartan 80 mg and HCTZ (Hydrochlorothiazide) and/or any other therapies commonly used in the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have met the inclusion criteria for the preceding clinical trial of telmisartan. All patients must give a separate written informed consent for participation in the open-label follow-up.

  * Mild-to-moderate essential hypertension defined as a mean seated diastolic blood pressure measurement of ≥ 95 mmHg measured by manual cuff sphygmomanometer
  * Mean seated systolic blood pressure ≥ 140 mmHg, measured my manual cuff
  * A 24-hour mean diastolic blood pressure, measured by ABPM (ambulatory blood pressure measurement), of ≥ 85 mmHg
  * Age 18 or older
  * Patient's written informed consent in accordance with GCP (Good Clinical Practice) and local legislation

Exclusion Criteria:

* Patients with a clinically significant change in ECG from baseline that was reported as an adverse event during the preceding clinical trial
* Patients who have developed a medical condition during the preceding clinical trial that, in the investigator's opinion, may be worsened by treatment or may compromise the safety evaluation of telmisartan
* Patients who discontinued the preceding telmisartan clinical trial due to an adverse event
* Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 1998-06; Primary Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Achievement of goal blood pressure response defined by a mean sitting diastolic blood pressure <90 mmHg | Up to one year
Need for addition of hydrochlorothiazide or subsequent change in antihypertensive therapy | Up to one year
Time to addition of hydrochlorothiazide or any subsequent change in antihypertensive therapy | Up to one year
Mean sitting diastolic blood pressure during each visit | At months 3, 6, 9, 12
Mean sitting systolic blood pressure during each visit | At months 3, 6, 9, 12
Number of patient with adverse events | Up to one year
Changes from baseline in heart rate | Baseline and at months 3, 6, 9, 12
Number of patients with abnormal changes in 12-Lead ECG (electrocardiogram) | Baseline and 12 months
Number of patients with abnormal changes in laboratory parameters | Baseline and 12 months
Number of patients with abnormal findings in physical examination | Baseline and at 12 month